CLINICAL TRIAL: NCT04411381
Title: Telemedicine-based Model of Care for the Management of Hepatitis C Infected Patients: a Randomized Clinical Trial
Brief Title: Telemedicine-based Model of Care for the Management of Hepatitis C Infected Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of La Laguna (Other)
Responsible Party: Principal Investigator, Manuel Hernandez-Guerra, MD, Head of Gastroenterology and Hepatology, University of La Laguna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TELE_RVS
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Hepatitis C; Telemedicine
MeSH Terms: conditions — Hepatitis C | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine-based model of care (Active Comparator): Telemedicine associated with dried blood spot testing at home for RNA test to sustained virological response determination
  Interventions: Other: Telemedicine
- Traditional model of care (No Intervention): Tradiotional model of care with venipuncture for RNA test to sustained virological response determination and face-to-face consultation

INTERVENTIONS:
Other: Telemedicine — Telemedicine associated with dried blood spot testing at home for RNA test to sustained virological response determination
  Arms: Telemedicine-based model of care

SUMMARY:
To achieve World Health Organization 2030 goals of hepatitis C elimination it is mandatory to document after treatment sustained virological response (SVR). Currently, patients after completing treatment do not show up for SVR assessment. The main objective of this study is to evaluate the effectiveness of a telemedicine-based model of care associated with dried blood spot testing at home to assess hepatitis C sustained virological response after treatment compared to the traditional model of care.

DETAILED DESCRIPTION:
This is a prospective, randomized study in which hepatitis C (VHC) infected patients will be randomized to two strategies for HCV care.

All HCV infected patients will be evaluated in a first face-to-face consultation with the hepatologist for fibrosis evaluation and treatment prescription the same day. Patients will be invited to participate if they are: 1) 18 years or older 2) have contact telephone number 3) sing the informed consent 4) have not advanced fibrosis (F3) or cirrhosis (F4) 5) are not under surveillance by another specialist or drug addiction centre.

Participants will be randomized into two strategies to assess sustained virological response (SVR) during follow-up:

1. The traditional model of care: one appointment for venipuncture for RNA testing to assess SVR (undetectable RNA 12 weeks after treatment cessation), and an appointment with the specialist for result communication.
2. Telemedicine-based model of care: The patient will be provided with a home kit to perform the dried blood spot (DBS) testing for HCV RNA at 12 weeks (SVR), and an appointment for teleconsultation and communicate the results.

Demographic, clinical and laboratory data will be collected to evaluate the characteristics of included patients and to study predictive factors of adherence.

A satisfaction questionnaire will be conducted to compare patients´ satisfaction with both health care models.

The hypothesis of the study is that the adherence and SVR determination record will increase using the telemedicine-based model of care.

For the present study, a 20% improvement in the adherence (SVR record) was hypothesized in the group of patients randomized to the telemedicine-based model of care compared to the traditional model of care. Taking into account power of 80%, alpha error of 5% and losses of 10% will require 68 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* have contact telephone number
* sing the informed consent

Exclusion Criteria:

* have advanced fibrosis (F3) or cirrhosis (F4)
* are under surveillance by another specialist or drug addition center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the two models of care | 12 months
  SVR record rate

SECONDARY OUTCOMES:
Acceptance of the intervention with a validated satisfaction questionnaire | 12 months
  Grade of patient satisfaction with telemedicine by a validated questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa CRUZ DE Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gomez L, Reygosa C, Morales-Arraez DE, Ramos R, Perez A, Hernandez A, Quintero E, Gutierrez F, Diaz-Flores F, Hernandez-Guerra M. Diagnostic test accuracy of the cobas 6800 system for detection of hepatitis c virus viraemia levels from dried blood spots. Enferm Infecc Microbiol Clin (Engl Ed). 2020 Jun-Jul;38(6):267-274. doi: 10.1016/j.eimc.2019.10.009. Epub 2019 Dec 4. English, Spanish. PMID 31812456
- [Background] Averhoff F, Shadaker S, Gamkrelidze A, Kuchuloria T, Gvinjilia L, Getia V, Sergeenko D, Butsashvili M, Tsertsvadze T, Sharvadze L, Zarkua J, Skaggs B, Nasrullah M. Progress and challenges of a pioneering hepatitis C elimination program in the country of Georgia. J Hepatol. 2020 Apr;72(4):680-687. doi: 10.1016/j.jhep.2019.11.019. Epub 2019 Dec 4. PMID 31811882
- [Background] Cuadrado A, Llerena S, Cobo C, Pallas JR, Mateo M, Cabezas J, Fortea JI, Alvarez S, Pellon R, Crespo J, Echevarria S, Ayesa R, Setien E, Lopez-Hoyos M, Crespo-Facorro B, Aguero J, Chueca N, Garcia F, Calleja JL, Crespo J. Microenvironment Eradication of Hepatitis C: A Novel Treatment Paradigm. Am J Gastroenterol. 2018 Nov;113(11):1639-1648. doi: 10.1038/s41395-018-0157-x. Epub 2018 Jun 27. PMID 29946175
- [Background] Jimenez Galan G, Alia Alia C, Vegue Gonzalez M, Garcia Berriguete RM feminine, Fernandez Gonzalez F, Fernandez Rodriguez CM, Gonzalez Fernandez M, Gutierrez Garcia ML, Losa JE, Velasco M, Moreno L, Hervas R, Delgado-Iribarren A, Palacios Garcia-Cervigon G. The contribution of telemedicine to hepatitis C elimination in a correctional facility. Rev Esp Enferm Dig. 2019 Jul;111(7):550-555. doi: 10.17235/reed.2019.6152/2018. PMID 31215210